CLINICAL TRIAL: NCT03109067
Title: Influence of TaqIB (rs708272) Polymorphism in Cholesteryl Ester Transfer Protein (CETP) Gene on Functionality of HDL Particles, in the Pathway of Reverse Transport of Fasting and Post-prandial Cholesterol.
Brief Title: Genetic and Metabolism of Post-prandial HDL Particles
Acronym: HDL-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: C10-57
Record Dates: First submitted 2017-03-01; First posted 2017-04-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Cholesterol, HDL, Postprandial Period, Polymorphism, Genetic

STUDY DESIGN:
Intervention Model Description: Same intervention for everyone, two different groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standardized meal (Experimental): Standardized meal for :
  50 patients with a TaqIB AA polymorphism 50 patients with a TaqIB GG polymorphism
  Interventions: Other: Standardized meal

INTERVENTIONS:
Other: Standardized meal — Blood samples performed at 5 different times : H0 before the meal, H2, H4, H6 and H8 after the meal

SUMMARY:
Reverse cholesterol transport (RCT) pathway explains the anti-atherosclerosis role of HDL. Post prandial hypertriglyceridemia is highly predictive of atherosclerosis. TaqIB polymorphism in CETP gene plays a role on HDL particles, and might give a link between TaqIB polymorphism and the cardioprotective efficiency of HDL particles. Our main objective was to compare post-prandial HDL particles between patients having B2 allele carriers (genotype AA) to B1 allele carriers (genotype GG), and their ability to mediate cellular cholesterol efflux, via SR-BI Scavenger Receptor class B type I (SR-BI) , ABCG1 and ABCA1 pathways.

DETAILED DESCRIPTION:
Background:

This trial focuses on anti-atherogenic properties functions of HDL lipoproteins, particularly those linked to reverse transport cholesterol (RCT) pathway, genetic factors involved in plasmatic HDL-C and post-prandial metabolism. The post-prandial period is associated with an activation of the RCT with an increase in Cholesteryl ester transfer protein (CETP), in plasmatic HDL particles. There is also an increase of HDL particles ability to mediate cellular cholesterol efflux, via SR-BI and ABCG1 pathways. TaqIB polymorphism is associated with a variation of the plasma to mediate cellular cholesterol efflux.

Aim of the study:

The investigators were aiming to test the hypothesis that the genetic variability of HDL-C is associated with structural and functional variability of post-prandial HDL particles and particularly in their ability to mediate the initial step of RCT.

Intervention:

The study aimed to include n=50 patients with a TaqIB AA polymorphism and 50 patients with a GG TaqIB polymorphism. Blood samples were performed fasted, before and after intake of a standardized test meal at 5 different time : H0 before the meal, H2, H4, H6 and H8 after the meal.

Explorations:

For the fasted sample a full lipidic assessment was performed including the dosing of: triglyceridemia, HDL-C, apolipoprotein B (apoB), apolipoprotein AI. The plasmatic kinetic of triglyceridemia, apoB100, apo-48 and the activity of CETP was performed on each sample.

HDL particles were also explored with qualitative and quantitative assessment of the HDL fractions ability to mediate cholesterol efflux via each pathway : SR-BI, ABCA1 and ABCG1 in our cellular models.

The study therefore aimed to improve our knowledge of molecular mechanisms involved in HDL particles dysfunction in metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Affiliation to a national social security scheme
2. Age between 18 and 60 years old
3. Male subjects
4. Participants harboring either a B2 (genotype AA) allele or a B1 (genotype GG) in TaqIB polymorphism of CETP gene
5. Fasted plasmatic triglyceridemia < 300 mg/dL
6. Free prior and informed written consent given by the participant

Exclusion Criteria:

1. Participants with an history of symptomatic cardio-vascular disease (infarct, angina pectoris, acute coronary syndrome, cardiac surgery, endoluminal coronal intervention, stroke, symptomatic peripheral artery disease) within 6 months prior to inclusion.
2. Triglyceridemia > 3 g/L
3. Participants having other lipid-lowering agents than statin (fibrate, niacin, ezetimibe)
4. Participants having a treatment (either systemic or local) which might interfere with the evaluation of study parameters.
5. Excessive alcohol consumption, or any drug addiction. An excessive alcohol consumption is superior to 21 time 30 mL of alcohol or 120 mL of wine or 355 mL of beer.
6. Regular smoker or smoking cessation within the last year
7. Significant abnormality on the full blood count or plasmatic and urinary biochemistry analysis.
8. Chronic or acute disease either life threatening or able to modify study results, including among others :

   1. Diabetes
   2. Renal diseases : nephrotic syndrome, chronic kidney failure and/or creatininemia > 1.7 time the upper limit of normal (ULN).
   3. Hypothyroidism defined by thyroid-stimulating hormone > 2x ULN
   4. Hepatobiliary disease or viral hepatitis B or C confirmed by transaminases > 2x ULN or alkaline phosphatase > 1.5x ULN or total bilirubinemia > 1.5x ULN at screening.
   5. Known HIV
   6. Gastro-intestinal disorder or disease that might modify intestinal absorption, bariatric surgery.
9. Participant who might interfere with the quality of the study or might compromise the study according to the investigator.
10. Participant currently enrolled in another study or in the exclusion period of another study.
11. Participants with uncontrolled hypertension defined by a systolic blood pressure > 140 mmHg or a diastolic blood pressure > 90 mmHg.
12. Participants with a C reactive protein (CRP) > 5mg/L
13. Participants with a E2/E2 phenotype of apolipoprotein E.
14. Blood donation or product derived-from blood donation within the last 3 months prior to the test meal.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2015-11-21 (Actual); Study Completion 2015-11-21 (Actual)

PRIMARY OUTCOMES:
Comparison of post-prandial HDL particles | before the meal (time = 0 hour) vs 2 hours after
  Compare post-prandial HDL particles area under curve (AUC) between patients having B2 allele carriers (genotype AA) to B1 allele carriers (genotype GG)

SECONDARY OUTCOMES:
Comparison of post-prandial HDL particles | before the meal (time = 0 hour), 2 hours, 4 hours, 6 hours and 8 hours after the meal
  Compare post-prandial HDL particles area under curve (AUC) between patients having B2 allele carriers (genotype AA) to B1 allele carriers (genotype GG), and their ability to mediate cellular cholesterol efflux, via SR-BI, ABCG1 and ABCA1 pathways.
Efflux capacity of postprandial HDL particles | before the meal (time = 0 hour), 2 hours, 4 hours, 6 hours and 8 hours after the meal
  - Compare the increase of efflux capacity of postprandial HDL particles between individuals harboring a B2 allele compared to those harboring a B1 allele.
Area under curves of triglyceridemia of apoB100 and apoB48 | before the meal (time = 0 hour), 2 hours, 4 hours, 6 hours and 8 hours after the meal
  Compare area under curves of triglyceridemia of apoB100 and apoB48 between individuals harboring a B2 allele (genotype AA) in the TaqIB polymorphism of the CETP gene.
Plasmatic concentrations of apoB100 | before the meal (time = 0 hour), 2 hours, 4 hours, 6 hours and 8 hours after the meal
  Compare plasmatic concentrations of apoB100 between individuals harboring a B2 allele (genotype AA) in the TaqIB polymorphism of the CETP gene.
Correlation between the area under curve of triglyceridemia and the efflux capacity of HDL particles. | before the meal (time = 0 hour), 2 hours, 4 hours, 6 hours and 8 hours after the meal
  Investigate the correlation between the area under curve of triglyceridemia and the efflux capacity of HDL particles.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ammour, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre d'Investigation Clinique Paris Est, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamaziere A, Rainteau D, Kc P, Humbert L, Gauliard E, Ichou F, Ponnaiah M, Bouby N, Salem JE, Mallet JM, Guerin M, Lesnik P. Distinct Postprandial Bile Acids Responses to a High-Calorie Diet in Men Volunteers Underscore Metabolically Healthy and Unhealthy Phenotypes. Nutrients. 2020 Nov 19;12(11):3545. doi: 10.3390/nu12113545. PMID 33228154
- [Background] Motte AM, Gall JG, Salem JE, Dasque E, Lebot M, Frisdal E, Galier S, Villard EF, Bouaziz-Amar E, Lacorte JM, Charbit B, Le Goff W, Lesnik P, Guerin M. Reduced Reverse Cholesterol Transport Efficacy in Healthy Men with Undesirable Postprandial Triglyceride Response. Biomolecules. 2020 May 25;10(5):810. doi: 10.3390/biom10050810. PMID 32466286
- [Background] Galier S, Darabi M, Ma F, Materne C, Guillas I, Le Goff W, Kontush A, Guerin M. Reduced Capacity of High-Density Lipoprotein to Acquire Free Cholesterol From Triglyceride-Rich Lipoproteins Is Associated With Elevated Postprandial Hypertriglyceridemia in Healthy Men. J Am Heart Assoc. 2024 Aug 6;13(15):e034770. doi: 10.1161/JAHA.123.034770. Epub 2024 Jul 31. PMID 39082393